CLINICAL TRIAL: NCT03500822
Title: Effects of Dynamic Hyperinflation on the Left-ventricular Diastolic Function in Healthy Male Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Otto Wagner Hospital (Other)
Responsible Party: Principal Investigator, Georg-Christian Funk, Head of Intensive Care Unit, Principal Investigator, Otto Wagner Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: Hyperstolic-COPD
Record Dates: First submitted 2018-02-09; First posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: dynamic hyperinflation; diastolic dysfunction; COPD; Chronic Obstructive Pulmonary Disease; Metronome-paced Tachypnea; Expiratory-stenosis Breathing
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Metronome-paced tachypnea (Experimental): Dynamic hyperinflation by the method of metronome-paced tachypnea.
  Interventions: Procedure: Metronome-paced tachypnea
- Exspiratory-stenosis breathing (Experimental): Dynamic hyperinflation by the method of expiratory-stenosis breathing.
  Interventions: Procedure: Expiratory-stenosis breathing

INTERVENTIONS:
Procedure: Metronome-paced tachypnea — three cycles: breathing frequency (BF) - 40/min, inspiration : expiration (I : E) - 1 : 1; BF - 40/min, I : E - 1 : 2; BF - 30/min, I : E - 1 : 2
  Other Names: MPT
  Arms: Metronome-paced tachypnea
Procedure: Expiratory-stenosis breathing — three cycles: BF - /min, I : E - 1 : 3; stenosis: 3mm; 2mm; 1,5mm
  Other Names: ESB
  Arms: Exspiratory-stenosis breathing

SUMMARY:
The aim of this study is to identify whether actively induced dynamic hyperinflation can cause left-ventricular diastolic dysfunction in healthy male subjects in order to explore the mechanisms of developing cardiac dysfunctions in patients with COPD.

DETAILED DESCRIPTION:
Cardiovascular diseases, especially left-ventricular diastolic dysfunction, are among the most frequent reasons for morbidity and mortality in patients with chronic obstructive pulmonary disease (COPD).

Dynamic hyperinflation is one of the expected pathophysiological mechanisms in the multifactorial genesis of this left-ventricular diastolic dysfunction in patients with COPD.

The novel concept of Expiratory Stenosis Breathing (ESB) is based on the method of Metronome-Paced Tachypnea (MPT) of Cooper et al. Therefore the investigators use a metronome to indicate a specific breathing frequency (BF) and the relation of inspiration : expiration (I : E) in order to let subjects hyperinflate.

Subjects get split into two groups each hyperinflating three times for 90sec by one of the two methods before doing a cross-over and switch groups to do the same in the other group. At the end of the 90sec there is a measurement of the Inspiratory Capacity (IC) and an echocardiography in order to objectify dynamic hyperinflation respectively the change in diastolic function.

During ESB participants hyperinflate with a BF - 30/min and a I : E - 1 : 3. In addition they have to breathe through an expiratory-effective stenosis (3, 2 and 1,5mm) on the mouthpiece of the pneumotachograph to simulate the collapsing airways in COPD-patients. In contrast, during MPT subjects hyperinflate with a BF - 40/min, I : E - 1 : 1; BF - 40/min, I : E - 1 : 2; BF - 30/min, I : E - 1 : 2.

During the whole trial investigators measure Intrinsic Positive Endexpiratory Pressure (PEEPi) in order to objectify the dynamic hyperinflation more significantly.

The primary goal of this study is to assess if actively induced dynamic hyperinflation can affect diastolic function of the left ventricle.

Furthermore a correlation between the extent of dynamic hyperinflation and diastolic dysfunction should be quantified.

In addition measurement of PEEPi should validate the method of Metronome-paced Tachypnea (MPT) because the investigators hypothesize that this method does not simulate the pathophysiological circumstances in patients with COPD sufficiently.

ELIGIBILITY:
Inclusion Criteria:

* BMI <27 kg/m2
* Lifelong nonsmoker (currently non-smoking and up to now less than 100 cigarettes)

Exclusion Criteria:

* Obstructive pulmonary diseases (asthma, COPD)
* Cardiovascular diseases (cardiac insufficiency, coronary heart diseases, hypertonia)
* Other relevant pulmonary or cardiac diseases
* Baseline E/A-ratio <1

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2016-11; Primary Completion 2017-09 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
E/A-ratio (absolute change between tidal breathing and smallest stenosis) | At the end of each cycle - tidal breathing as well as hyperinflation-intervention (each cycle is at least 90 seconds).
  E/A-ratio will be measured by transthoracic echocardiography (Vivid S9, general electric healthcare, Fairfield, USA) according to the valid standards of The European Association of Echocardiography. This parameter represents the left-ventricular diastolic function.

SECONDARY OUTCOMES:
E/E'-ratio | At the end of each cycle - tidal breathing as well as hyperinflation-intervention (each cycle is at least 90 seconds).
  E/E'-ratio will be measured by transthoracic echocardiography (Vivid S9, general electric healthcare, Fairfield, USA) according to the valid standards of The European Association of Echocardiography. This parameter represents the left-ventricular diastolic function.
deceleration time of the E-wave transmitral (msec) | At the end of each cycle - tidal breathing as well as hyperinflation-intervention (each cycle is at least 90 seconds).
  deceleration time will be measured by transthoracic echocardiography (Vivid S9, general electric healthcare, Fairfield, USA) according to the valid standards of The European Association of Echocardiography. This parameter represents the left-ventricular diastolic function.
Maximal diastolic transtricuspid flow (m/sec) | At the end of each cycle - tidal breathing as well as hyperinflation-intervention (each cycle is at least 90 seconds).
  Maximal diastolic transtricuspid flow will be measured by transthoracic echocardiography (Vivid S9, general electric healthcare, Fairfield, USA) according to the valid standards of The European Association of Echocardiography. This parameter represents the left-ventricular diastolic function.
Maximal late-systolic velocity of the lateral tricuspid valve in Tissue Doppler Imaging (cm/sec) | At the end of each cycle - tidal breathing as well as hyperinflation-intervention (each cycle is at least 90 seconds).
  Maximal late-systolic velocity will be measured by transthoracic echocardiography (Vivid S9, general electric healthcare, Fairfield, USA) according to the valid standards of The European Association of Echocardiography. This parameter represents the left-ventricular diastolic function.
Inspiratory Capacity | At the end of each cycle - tidal breathing as well as hyperinflation-intervention (each cycle is at least 90 seconds).
  Inspiratory Capacity will be measured with a pneumotachograph (VenThor D-22/5B, ThorMedical, Budapest, Hungary). It represents the extent of dynamic hyperinflation.
Dynamic Intrinsic Positive Endexpiratory Pressure: | During each entire cycle - tidal breathing as well as hyperinflation-intervention (each cycle is at least 90 seconds).
  To objectify the dynamic hyperinflation in addition to the Inspiratory Capacity, the Intrinsic Positive Endexpiratory Pressure will be measured by the invasive application of an esophageal balloon catheter (ICU-Lab, Kleistek Engineering, Bari, Italy).

CONTACTS AND LOCATIONS:
Overall Officials: Georg C Funk, Assoc. Prof., Principal Investigator — Department of Respiratory and Critical Care Medicine and Ludwig-Boltzmann Institute for COPD and Respiratory Epidemiology, Otto Wagner Hospital, Vienna
Locations (1):
- Otto Wagner Spital, Dep. of Respiratory and Critical Care Medicine, Vienna, Austria

REFERENCES:
- [Background] Cooper CB, Calligaro GL, Quinn MM, Eshaghian P, Coskun F, Abrazado M, Bateman ED, Raine RI. Determinants of dynamic hyperinflation during metronome-paced tachypnea in COPD and normal subjects. Respir Physiol Neurobiol. 2014 Jan 1;190:76-80. doi: 10.1016/j.resp.2013.08.002. Epub 2013 Aug 27. PMID 23994176
- [Background] Weigt SS, Abrazado M, Kleerup EC, Tashkin DP, Cooper CB. Time course and degree of hyperinflation with metronome-paced tachypnea in COPD patients. COPD. 2008 Oct;5(5):298-304. doi: 10.1080/15412550802363428. PMID 18972278
- [Background] Evangelista A, Flachskampf F, Lancellotti P, Badano L, Aguilar R, Monaghan M, Zamorano J, Nihoyannopoulos P; European Association of Echocardiography. European Association of Echocardiography recommendations for standardization of performance, digital storage and reporting of echocardiographic studies. Eur J Echocardiogr. 2008 Jul;9(4):438-48. doi: 10.1093/ejechocard/jen174. PMID 18579482
- [Background] Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, Crapo R, Enright P, van der Grinten CP, Gustafsson P, Jensen R, Johnson DC, MacIntyre N, McKay R, Navajas D, Pedersen OF, Pellegrino R, Viegi G, Wanger J; ATS/ERS Task Force. Standardisation of spirometry. Eur Respir J. 2005 Aug;26(2):319-38. doi: 10.1183/09031936.05.00034805. No abstract available. PMID 16055882
- [Background] Akoumianaki E, Maggiore SM, Valenza F, Bellani G, Jubran A, Loring SH, Pelosi P, Talmor D, Grasso S, Chiumello D, Guerin C, Patroniti N, Ranieri VM, Gattinoni L, Nava S, Terragni PP, Pesenti A, Tobin M, Mancebo J, Brochard L; PLUG Working Group (Acute Respiratory Failure Section of the European Society of Intensive Care Medicine). The application of esophageal pressure measurement in patients with respiratory failure. Am J Respir Crit Care Med. 2014 Mar 1;189(5):520-31. doi: 10.1164/rccm.201312-2193CI. PMID 24467647
- [Background] Anthonisen NR, Connett JE, Enright PL, Manfreda J; Lung Health Study Research Group. Hospitalizations and mortality in the Lung Health Study. Am J Respir Crit Care Med. 2002 Aug 1;166(3):333-9. doi: 10.1164/rccm.2110093. PMID 12153966
- [Background] Lopez-Sanchez M, Munoz-Esquerre M, Huertas D, Gonzalez-Costello J, Ribas J, Manresa F, Dorca J, Santos S. High Prevalence of Left Ventricle Diastolic Dysfunction in Severe COPD Associated with A Low Exercise Capacity: A Cross-Sectional Study. PLoS One. 2013 Jun 27;8(6):e68034. doi: 10.1371/journal.pone.0068034. Print 2013. PMID 23826360
- [Background] Barr RG, Bluemke DA, Ahmed FS, Carr JJ, Enright PL, Hoffman EA, Jiang R, Kawut SM, Kronmal RA, Lima JA, Shahar E, Smith LJ, Watson KE. Percent emphysema, airflow obstruction, and impaired left ventricular filling. N Engl J Med. 2010 Jan 21;362(3):217-27. doi: 10.1056/NEJMoa0808836. PMID 20089972
- [Derived] Urban MH, Mayr AK, Schmidt I, Grasmuk-Siegl E, Burghuber OC, Funk GC. Effects of Dynamic Hyperinflation on Left Ventricular Diastolic Function in Healthy Subjects - A Randomized Controlled Crossover Trial. Front Med (Lausanne). 2021 May 4;8:659108. doi: 10.3389/fmed.2021.659108. eCollection 2021. PMID 34017848